CLINICAL TRIAL: NCT05349487
Title: Evaluation of a Disposable Hands-Free Heat and Moisture Exchanger (HME) Valve: The Blom-Singer SpeakFree HME Hands Free Valve
Brief Title: SpeakFree Heat and Moisture Exchanger (HME)
Acronym: SPEAKFREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mario Alberto Landera, SLP.D, Associate Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20210501
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Laryngeal Cancer; Laryngectomy
Keywords: Stoma; Voice Prosthesis; Total Laryngectomy; Heat and Moisture Exchanger (HME)
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SpeakFree Hands Free Heat Moisture Exchanger (HEM) Valve Group (Experimental): Participants will be fitted to use a hand free HME device over their stoma in order to communicate with a voice prosthesis for one month. The participants will also serve as their own control performing voicing and speech tasks using digital occlusion and digital depression HME.
  Interventions: Device: SpeakFree HME Hands Free Valve; Other: Digital Occlusion; Device: Digital Depression HME

INTERVENTIONS:
Device: SpeakFree HME Hands Free Valve — A voice prosthesis, SpeakFree HME Hands Free Valve, achieved with creation of a tracheoesophageal puncture will be placed over the stoma for 1 month.
Other: Digital Occlusion — Using participant's own fingers, they will be putting their fingers over the stoma.
Device: Digital Depression HME — A digital handheld press-down HME will be placed over stoma.

SUMMARY:
The purpose of the study is to evaluate the new Blom-Singer SpeakFree disposable hands free valve heat and moisture exchanger (HME). The investigators will compare the SpeakFree to other modalities of stomal occlusion (digital occlusion and digital depression of an HME) for patients who communicate with a voice prosthesis as determined by patient preference and satisfaction. In addition, the investigators will compare the SpeakFree to other modalities of stomal occlusion as determined by objective measures of speech and voice parameters (maximum phonation time, syllables per breath, minimum/maximum phonation pressures, and a clinician rating of voice quality using a visual analog scale).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have undergone a total laryngectomy who have and use a voice prosthesis as their primary form of communication for at least 3 months prior to study enrollment.
* Participants must have had at least 2 voice prosthesis management visits from a speech pathologist at the University of Miami prior to study enrollment.
* Participants must have fully healed suture lines.
* Participants must demonstrate fluent tracheoesophageal speech (i.e., maximum phonation time of at least 5 seconds during 3 consecutive trials)
* Current HME use for a minimum of 1 month
* Participants willing to complete the survey and provide a signed Informed Consent Form
* Males and non-pregnant females over the age of 18

Exclusion Criteria:

* Participants who do not have a voice prosthesis.
* Participants who have dysarthria.
* Participants who are currently receiving treatment for head and neck cancer.
* Participants who have an underlying neurologic condition potentially impacting speech.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction as measured by VAS | Up to 1 month
  Patient preference and satisfaction will be measured using a visual Analog Scale (VAS) ranging in score from 1-10 with a higher score indicating greater satisfaction with the device.
Voice Quality: Patient Rating | Up to 1 month
  Voice Quality will be measured using a visual Analog Scale ranging in score from 1-10 with a higher score indicating that the patient feels their voice quality is better with the device.

SECONDARY OUTCOMES:
Change in Maximum Phonation Time | Baseline, 1 month
  Maximum phonation time (MPT) is a clinical measurement of the longest time a person can phonate a vowel in seconds.
Change in Syllables Per Breath | Baseline, 1 month
  Participants' number of syllables per breath while reading a standardized reading passage will be measured and reported.
Pressure Needed to Phonate | Baseline
  Minimal and maximal pressures will be reported using a manometer while the participant counts from 1 to 15.
Change in Voice Quality: Clinician Rating | Baseline, 1 month
  The clinician will rate participant's voice quality using VAS. VAS has a total score ranging from 1 to 10 with the higher score indicating that the clinician feels that participant's voice quality is better with the device.

CONTACTS AND LOCATIONS:
Overall Officials: Mario A Landera, SLP.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No